CLINICAL TRIAL: NCT04317638
Title: Lipid Profile of Full-term Infants on Different Feeding Regimen: a Comparative Study
Brief Title: Lipid Profile of Infants on Different Feeding Regimens
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maria Remon Riad Sedrak, Doctor, Assiut University
Other Study IDs: Lipid profile of infants
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Lipid Profile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- breastfed group: Infants on exclusive breast feeding for the first 6 months of life and their mothers
  Interventions: Other: Lipid profile
- formula fed group: Infants on exclusive formula feeding for the first 6 months of life
  Interventions: Other: Lipid profile
- mixed fed group: Infants on mixed feeding (formula & breast feeding) and their mothers
  Interventions: Other: Lipid profile

INTERVENTIONS:
Other: Lipid profile — 3 ml of venous blood from the breastfed and infants and mothers of the breastfed and mixed fed infants will be taken under aseptic precautions for determination of triglycerides (TG), cholesterol, high density lipoprotein (HDL), very low density lipoprotein (LDL) at the age of 14 ± 2 weeks and the age of 6 months.

SUMMARY:
Lipid profile of full-term infants on different regimens. The aim of the study is to compare infant's lipid profiles on different feeding regimen during the first 6 months of life and its correlation with their mothers' lipid profiles (exclusive breastfeeding and mixed feeding) and to compare infants' lipid profiles on different feeding regimen with each other (including those on exclusive formula feeding).

DETAILED DESCRIPTION:
Infant and young child feeding is critical for their health and survival. Based on well-established evidence, the World Health Organization (WHO) and the United Nations Children's fund (UNICEF) recommend that mothers put newborns to the breast within one hour of birth, breastfeed infants exclusively for the first six months and continue to breastfeed for two years and beyond, together with nutritionally adequate, safe, age-appropriate, responsive feeding of solid, semi-solid and soft food starting in the sixth month.

For the first six months of life, breast milk alone is the ideal nourishment, providing all of the nutrients including minerals and fat soluble vitamins, an infant needs, meaning that no other liquid or food is needed.

In addition to providing a generally adequate nutrient supply that support normal growth and development , breastfeeding has been linked to multiple other advantages including a reduced risk of infection and long-term benefits for the risk of obesity, type II diabetes mellitus, blood pressure and better performance in intelligence tests.

The macro-nutrient composition of human milk varies within mothers according to nutritional status and across lactation. The mean macro-nutrient composition of mature, term milk is estimated to be approximately 0.9 to 1.2 gm/dl for proteins, 3.2 to 3.6 gm/dl for fats and 6.7 to 7.8 gm/dl for lactose.

There have been several systematic reviews supporting the positive effects of breastfeeding on cardiovascular risk factors, such as obesity and type 2 diabetes (DMII), hypertension. Breastfeeding also reduces plasma levels of total cholesterol (TC) and low density lipoprotein (LDL).

Breast milk is a protective factor against obesity. This effect could be explained by existing differences in macro-nutrients. Moreover, there are physiological differences between breast milk and artificial formulas in terms of their nutrients and hormone contents. For instance, protein content of baby formulas is higher than that of breast milk, and leptin exists in breast milk, but not in artificial formulas. Due to their high fat and protein contents, baby formulas would lead to increased secretion of Insulin Growth Factor-type 1 (IGF-1),and subsequently to stimulation of adipocytes, which eventually result in excess weight. Moreover, breastfeeding affects the intake of calorie and protein, insulin secretion, balancing fat reserves, and adipocyte size. The effect of breastfeeding is found to be independent from dietary patterns and physical activity in adulthood.

Many studies have confirmed the protective role of breastfeeding against type II diabetes mellitus. This effect is considered to be because of the difference in composition of breast milk and the difference in hormones of insulin, motilin, introglucagon, neurotencin, and pancreatic polypeptide in breast milk and artificial formulas, which in turn would lead to lower subcutaneous fat deposition in breastfed infants.

The effect of breastfeeding on hypertension has attracted much interest because of the differences between breast milk and artificial formulas, mainly in terms of their content of sodium and fatty acids. It is documented that breastfeeding can affect systolic and diastolic blood pressures in adulthood. The effect of breastfeeding on blood pressure in adulthood can be partly explained through the following mechanisms: (1) reduced sodium intake in infancy, (2) high content of long-chain unsaturated fatty acids in breast milk, which is an important component of the tissue membrane system, as coronary endothelial system, (3) protection against hyperinsulinemia in infancy, as well as prevention of insulin resistance in early life, adolescence, and adulthood.

There is a relationship between the molecular composition (especially lipids, glycerides and sterols) of the maternal plasma, milk and her infant.

There is paucity of studies comparing lipid profiles of exclusively breastfed and mixed fed infants and those correlating lipid profiles of breastfed infants and their mothers' lipid profiles.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy infants during the first 6 months of life on different feeding regimen

Exclusion Criteria:

1. Infants with perinatal problems .e.g.,

   * birth asphyxia
   * premature rupture of membranes
   * hypoglycemia
   * hypothermia
   * meconium stained amniotic fluid
   * pathological jaundice
   * congenital malformations
   * clinical evidence of chromosomal abnormalities
2. Infants born to mothers having any chronic disease e.g.,

   * diabetes mellitus
   * gestational diabetes
   * hypertension
   * pre-eclampsia
   * eclampsia
   * hypo/hyperthyroidism
   * on any long-term medication

Ages: 12 Weeks to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants seeking medical advice in the outpatient clinics of Assiut University Children Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
comparison between lipid profiles of the infants of the 3 groups | baseline
  analysis of the results of lipid profiles of infants on different feeding regimens at the age of 14 weeks and 6 months
correlation of lipid profiles of infants and their mothers | baseline
  analysis of the results of lipid profiles of infants on exclusive breast feeding and mixed feeding (breast and formula feeding) and the results of lipid profiles of their mothers

CONTACTS AND LOCATIONS:
Overall Officials: Nagla H Abu Faddan, PHD, Study Chair — Assiut University Children Hospital; Amir M Abo El-Gheit, PHD, Study Chair — Assiut University Children Hospital

REFERENCES:
- [Background] Martin MA, Lassek WD, Gaulin SJ, Evans RW, Woo JG, Geraghty SR, Davidson BS, Morrow AL, Kaplan HS, Gurven MD. Fatty acid composition in the mature milk of Bolivian forager-horticulturalists: controlled comparisons with a US sample. Matern Child Nutr. 2012 Jul;8(3):404-18. doi: 10.1111/j.1740-8709.2012.00412.x. Epub 2012 May 24. PMID 22624983
- [Background] Harit D, Faridi MM, Aggarwal A, Sharma SB. Lipid profile of term infants on exclusive breastfeeding and mixed feeding: a comparative study. Eur J Clin Nutr. 2008 Feb;62(2):203-9. doi: 10.1038/sj.ejcn.1602692. Epub 2007 Feb 28. PMID 17327867
- [Background] Owen CG, Martin RM, Whincup PH, Smith GD, Cook DG. Does breastfeeding influence risk of type 2 diabetes in later life? A quantitative analysis of published evidence. Am J Clin Nutr. 2006 Nov;84(5):1043-54. doi: 10.1093/ajcn/84.5.1043. PMID 17093156